CLINICAL TRIAL: NCT00580398
Title: A Pilot Smoking Cessation Study for Newly Diagnosed Lung Cancer Patients
Brief Title: Smoking Cessation Intervention for Thoracic Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Elyse Park, PhD, Elyse Park, PhD, Principal Investigator, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007p-000838; 1R03CA130722-01 (NIH)
Record Dates: First submitted 2007-12-20; First posted 2007-12-24 (Estimated); Results first posted 2014-11-21 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2018-09

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Motivational Interviewing; Varenicline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Usual care included physician advice to quit smoking.
- Intervention (Experimental): Intervention participants were provided with a cognitive-behavioral 12-week program consisting of varenicline (1mg bid, with initial titration up over week 1) and smoking cessation counseling targeted to the issues of thoracic cancer patients. We offered 7 counseling sessions but were flexible in offering additional counseling when needed. Counseling was delivered by a certified Tobacco Treatment Counselor using Motivational Interviewing (MI) techniques.
  Interventions: Behavioral: Smoking cessation counseling; Drug: varenicline

INTERVENTIONS:
Behavioral: Smoking cessation counseling — Median of 9 tobacco treatment counseling sessions conducted in person or by telephone.
  Other Names: Motivational Interviewing
  Arms: Intervention
Drug: varenicline — varenicline (1mg bid, with initial titration up over week 1) for 12 weeks
  Other Names: Chantix
  Arms: Intervention

SUMMARY:
The primary aim of the proposed study is to develop and assess the feasibility of delivering a smoking cessation intervention to patients undergoing lung surgery that begins before surgery and continues up to 3 months post-discharge. The secondary aim is to assess smoking cessation rates 3 months following surgery.

DETAILED DESCRIPTION:
This is a pilot study evaluating the feasibility of a cognitive-behavioral smoking cessation plus Varenicline program, designed specifically for early stage lung cancer patients and patients with a potential lung cancer diagnosis pre and post-surgery. The study population will be approximately 80 smokers who have upcoming lung resection surgery scheduled at Massachusetts General Hospital (MGH) in Boston. A patient will be considered eligible for the intervention or control group if he or she 1) is scheduled for a lung resection surgery with either a lung cancer diagnosis or a potential lung cancer diagnosis, and 2) had a cigarette in the past 2 weeks, 3) is willing to make a pre-surgical quit attempt. Patients will be excluded from the control group if they are 1) non-English speaking, 2) determined medically ineligible by their surgeon/oncologist, 3) suffering from psychosis or dementia 4) is currently on Varenicline has been on Varenicline for more than 3 weeks, or 5) is otherwise unable to participate in the intervention. Patients will be excluded from the intervention group if they are 1) non-English speaking, 2) determined medically ineligible by their surgeon, 3) suffering from psychosis or dementia 4) have been taking Varenicline for longer than three weeks 5) have been taking Bupropion (for smoking cessation purposes) for more than three weeks, 6) is otherwise unable to participate in the intervention.

ELIGIBILITY:
Inclusion Criteria:

A patient is eligible if he/she:

1. Is scheduled for a lung resection surgery with either a lung cancer diagnosis or a potential lung cancer diagnosis
2. Smoked a cigarette in the past 2 weeks
3. Is willing to make a pre-surgical quit attempt

Exclusion Criteria:

Patients will be excluded from the intervention group if they are:

1. Non-English speaking
2. Determined medically ineligible by their surgeon
3. Suffering from psychosis or dementia
4. Have been taking Varenicline for longer than three weeks
5. Have been taking Bupropion (for smoking cessation purposes) for more than three weeks
6. Is otherwise unable to participate in the intervention.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2008-01; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elyse Park, Ph.D., Principal Investigator — MGH
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Result] Park ER, Japuntich S, Temel J, Lanuti M, Pandiscio J, Hilgenberg J, Davies D, Dresler C, Rigotti NA. A smoking cessation intervention for thoracic surgery and oncology clinics: a pilot trial. J Thorac Oncol. 2011 Jun;6(6):1059-65. doi: 10.1097/JTO.0b013e318215a4dc. PMID 21512406

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study used a non-randomized design, which began with a usual care control group enrollment period (January 2008-June 2008) that was followed by an intervention group (June 2008-August 2009)enrollment period. We recruited patients referred to thoracic surgery and oncology clinics at the Massachusetts General Hospital (MGH) in Boston, MA.
Pre-assignment Details: A patient had to be willing to take varenicline in order to be eligible for the intervention group; if a patient who was otherwise eligible for the intervention group was taking nicotine replacement therapy or bupropion, he/she had to be willing switch to varenicline.
Groups:
- Intervention: Intervention participants were provided with a 12-week program consisting of varenicline (1mg bid, with initial titration up over week 1) and smoking cessation counseling targeted to the issues of thoracic cancer patients. We had proposed to offer 7 counseling sessions but were flexible in offering additional sessions when needed. The counseling was delivered by a certified Tobacco Treatment Counselor using motivational interviewing (MI) techniques.
Period: Overall Study
Arm/Group | Control | Intervention
Started | 17 | 32
Completed | 17 | 32
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Intervention: 12-week program consisting of varenicline (1mg bid, with initial titration up over week 1) and smoking cessation counseling sessions targeted to the issues of thoracic cancer patients.
- Total: Total of all reporting groups
Arm/Group | Control | Intervention | Total
Number analyzed (Participants) | 17 | 32 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.0 (10.5) | 57.5 (13.4) | 57.7 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 20 | 29
  Male | 8 | 12 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 16 | 31 | 47
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 17 | 28 | 45
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Determination of the Feasibility of a Cognitive Behavioral Smoking Cessation Intervention.
Description: Number of participants who completed the 12-week follow-up survey and thus the study.
Time Frame: 12 weeks
Measure: Number; unit: participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 17 | 32
participants | 17 | 32

2. Secondary Outcome: Biochemically-validated 7-day Point Prevalence Tobacco Abstinence
Description: 7-day point prevalence abstinence ("Have you smoked a cigarette, even a puff, in the past 7 days?") was assessed at 12-week follow-up. Self reported abstinence was confirmed only if a salivary cotinine level was < 15 ng/ml or an expired carbon monoxide measurement was <10 ppm.
Time Frame: 12 weeks
Population: 46 participants (32 intervention, 14 control) returned a cotinine confirmation kit for biochemical validation of 7 day point prevalent tobacco abstinence at 12 weeks. 3 control participants were excluded from the follow-up analysis.
Measure: Number; unit: participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 14 | 32
participants | 2 | 11

ADVERSE EVENTS:
Time Frame: 2 years (duration of study)
Arm/Group | Control | Intervention
Serious Adverse Events (participants affected / at risk) | 0/17 | 1/32
Other Adverse Events (participants affected / at risk) | 0/17 | 0/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=17) | Intervention (N=32)
Psychiatric Instability (Psychiatric disorders) | 0 (0) | 1 (1) — Patient admitted for psychiatric evaluation for anxiety. At admission, patient was taking varenicline for 6 weeks per study protocol. Because varenicline can cause psychiatric side effects, event reported as possibly related to study medication.

LIMITATIONS AND CAVEATS:
The generalizability of the findings are limited by a single study site. The statistical power to detect differences was limited by the small sample size of this pilot study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No